CLINICAL TRIAL: NCT01512186
Title: A Phase II Study Investigating Upfront Pazopanib In Metastatic Clear Cell Renal Cancer (Panther)
Brief Title: A Phase II Study Investigating Upfront Pazopanib In Metastatic Renal Cancer Renal Cancer (Panther)
Acronym: Panther
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Queen Mary University of London (Other)
Responsible Party: Principal Investigator, Centre of Experimental Medicine, Thomas Powles, Queen Mary University of London
Other Study IDs: 2009-016675-29
Record Dates: First submitted 2011-10-04; First posted 2012-01-19 (Estimated); Last update posted 2014-06-12 (Estimated); Status verified 2014-06

CONDITIONS: Metastatic Clear Cell Renal Cancer
Keywords: Clear cell renal cancer

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Pre-treatment biopsy and post treatment nephrectomy samples will be obtained
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The purpose of this study is to investigate if 14 weeks of pazopanib therapy prior to surgery (nephrectomy) is of benefit to patients with metastatic renal cancer. Ninety-five patients will be recruited into his study.

DETAILED DESCRIPTION:
This is a Phase II, open label study evaluating pre-operative pazopanib treatment in previously untreated patients with metastatic clear cell renal cancer. This study follows a Simon 2 stage design

Patients will take pazopanib for 14 weeks followed by a nephrectomy. The drug will continue after nephrectomy until disease progression is documented. Patients will come off study once disease progression occurs, where they will then be followed for survival. Subsequent treatment at the discretion of the treating physician will be documented.

After surgery, all patients will be radiologically evaluated 8 weekly until progression. Standard radical nephrectomy with lymph node dissection will be performed on those patients who are deemed operable. The surgery can be laparoscopic or open. Those not deemed suitable for nephrectomy after 14 weeks of treatment will be offered a repeat biopsy.

ELIGIBILITY:
Inclusion Criteria:

* Histopathologically confirmed clear cell carcinoma with measurable metastases on CT/MRI imaging (by RECIST v1.1). Only a component of clear cell is required.

  * No prior systemic treatment or nephrectomy for RCC. Palliative radiotherapy is acceptable to non target lesions.
  * Adequate organ function as defined by the following criteria:

    i. Total serum bilirubin ≤1.5 x uln (patients with gilbert's disease exempt) ii. Serum transaminases (ALT) <3 x uln iii. Calculated creatinine clearance >30ml/min iv. Absolute neutrophil count (ANC) ≥1000/mm3 without growth factor support v. Platelets ≥ 75,000/mm3
  * Signed and dated informed consent document indicating that the patient (or legally acceptable representative) has been informed of all the pertinent aspects of the trial prior to enrolment.
  * Willingness and ability to comply with scheduled visits, treatment plans and laboratory tests and other study procedures
  * ECOG performance status of 0, 1 or 2.
  * 18 years or above (no upper age limit) Male or female

Exclusion Criteria:

* Congestive heart failure (class III or IV NYHA), myocardial infarction or coronary artery bypass graft/ stenting or stroke in the previous six months, ongoing severe or unstable arrhythmia requiring medication.

  * Previous treatment for renal cancer
  * Pregnancy or breastfeeding. Female patients must be surgically sterile, be postmenopausal, or must agree to use adequate contraception during the period of therapy.
  * Male patients must be surgically sterile or agree to use adequate contraception during the period of therapy.
  * Other severe acute or chronic medical or psychiatric condition, or laboratory abnormality that would in the judgement of the investigator, impart excess risk associated with study participation or study drug administration, or which, in the judgement of the investigator, would make the patient inappropriate for entry into this study
  * Prolonged QT interval >480msecs or a history of prolonged QT interval >480msecs
  * Ongoing major gastrointestinal disease including ulcerative colitis, bleeding peptic ulcer disease or inflammatory bowel disease.
  * Bleeding diathesis
  * Current uncontrolled hypertension
  * Another malignancy requiring treatment within the last 5 years. Local prostate cancer not requiring hormone therapy or an asymptomatic raised PSA is acceptable.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population for this trial are patients with confirmed clear cell carcinoma with measurable metastases on CT/MRI imaging (by RECIST). Only a component of clear cell is required.
Sampling Method: Probability Sample
Enrollment: 95 (Estimated)
Dates: Start 2010-07; Primary Completion 2014-02 (Actual); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
Clinical benefit of 14 weeks of pre-operative pazopanib therapy, prior to nephrectomy using RECIST 1.1 criteria | Interim analysis after 34 patients have 12 weeks of treatment
  12 week CT scan will be compared to the baseline CT scan using RESIST criteria 1.1 to assess whether the patients have benefited from the upfront pazopanib treatment.

SECONDARY OUTCOMES:
Surgical complications (blood loss, post operative complications, hospital stay) | After the first 20 patients have had a nephrectomy
  Following surgery information regarding the quantity of blood loss, time the surgery took, length of hospital stay and whether there were any surgical complications will be recorded.
Overall Survival | After three years of study
  Overall survival will be measured from start of treatment to time of death.
Progression free survival | After all patients have progresssed
  Progression free survival will be measured from start of study treatment to time of disease progression.
Local response of primary tumour to pazopanib | After 12 weeks of study drug

CONTACTS AND LOCATIONS:
Locations (9):
- United Kingdom (9):
  - Basildon and Thurrock University Hospitals NHS Foundation Trust, Basildon
  - University Hospitals Coventry & Warwickshire NHS Trust, Coventry
  - The Beatson West of Scotland Cancer Centre, Glasgow
  - Barts and London Hospital NHS Trust, London
  - Oncology & Clinical Haematology Trials Unit, Royal Free Hospital, London
  - Oncology & Haematology Clinical Trials Unit, Guy's Hospital, London
  - Department of Oncology Oxford Cancer Centre, Oxford
  - Southampton General Hospital, Southampton
  - Southend University Hospital Trust, Southend